CLINICAL TRIAL: NCT05394467
Title: A Novel Approach to Examine the Adipose Cellular Kinetics of Lipedema
Brief Title: Adipose Cellular Kinetics of Lipedema
Acronym: LIPEDEMA
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Lipedema Foundation (Other)
Responsible Party: Principal Investigator, Ursula White, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2021-051
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Lipedema
Keywords: Adipose tissue; Lipedema; Subcutaneous abdominal; Subcutaneous femoral; Adipocyte; Adipose turnover; Adipose kinetics; Adipogenesis; Deuterium; Obesity
MeSH Terms: conditions — Lipedema; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lipedema: Women with diagnosed lipedema

SUMMARY:
Lipedema is characterized by an abnormal deposition of adipose tissue, resulting in fluid accumulation, limb enlargement, and pain. Lipedema is often misdiagnosed as simply obesity. A major challenge with diagnosis is the poorly understood biology underlying the disease. Limited studies suggest that the development of lipedema may involve adipocyte hypertrophy, increased commitment of adipose progenitor cells, hypoxia, adipocyte necrosis and macrophage recruitment. There remains an urgent need to investigate novel characteristics of adipose remodeling that may contribute to the pathogenesis of lipedema. The study investigators have reported quantitative measures of in vivo adipose kinetics using an 8-week incorporation of deuterium (administered as 2H2O) into the adipose tissue of women with obesity. The objective of this proposal is to utilize the metabolic 2H-labeling approach to measure, for the first time, in vivo adipocyte formation and triglyceride synthesis in the adipose tissue of participants with lipedema. Imaging approaches will provide a range of measurements to characterize the lipedema depots. The investigators hypothesize that lipedema adipose depots will have higher rates of adipocyte formation and triglyceride synthesis than both non-lipedema depots and those of women with traditional obesity. Lipedema may involve adipose tissue remodeling, characterized by adipocyte hypertrophy and increased commitment of preadipocytes and differentiation of adipocytes (adipogenesis), yielding an abundance of adipocytes with limited capacity to expand and accommodate lipid, resulting in hypoxia, macrophage recruitment, and local/systemic inflammation. Findings from this proposal will contribute to a better understanding of the pathogenesis of lipedema and may provide insight for the future development of therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤50 kg/m2
* Waist/hip ratio <0.86 (standing position)
* Clinical diagnosis of lipedema (mostly Stage 3 but Stage 2 will not be excluded)
* Willing to drink deuterated water (2H2O)

Exclusion Criteria:

* Have major organ disease (heart, kidney, lung, thyroid, liver) or abnormal liver enzymes that represent a problem for study inclusion
* Chronic use of systemic glucocorticoids, atypical anti-psychotic medications, or medications that cause clinically significant changes in weight
* Pregnancy or breastfeeding in the next 3 months
* Partial and/or full hysterectomy (due to estrogen effects on adipogenesis)
* PCOS
* Self-reported positive test for HIV, hepatitis B and hepatitis C
* Smoking or use of tobacco products in the last 6 months
* Any medical, psychiatric or behavioral factors that may interfere with study participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with diagnosed lipedema will be recruited and enrolled at Pennington Biomedical Research Center. A racially/ethnically diverse population will be recruited based on the local demographics
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess in vivo adipocyte formation in lipedema adipose depots (femoral) and non-lipedema depots (abdominal,) from patients with lipedema. | 8 weeks
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is enriched into the DNA of newly formed adipocytes. Lipedema adipose depots (femoral) will be compared to non-lipedema depots (abdominal) in these women with lipedema.

SECONDARY OUTCOMES:
Assess in vivo triglyceride formation in lipedema adipose depots (femoral) and non-lipedema depots (abdominal,) from patients with lipedema. | 8 weeks
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is enriched into the glycerol moiety of triglycerides, reflecting recent triglyceride formation. Lipedema adipose depots (femoral) will be compared to non-lipedema depots (abdominal) in these women with lipedema.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No